CLINICAL TRIAL: NCT05395676
Title: The Effect of Cognitive Exergame Training on Dual-Task Cost and Balance Stability of the Individuals Between 65 and 85 Years
Brief Title: Cognitive Exergame Training on Dual-Task Cost and Balance Stability in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Ahmet Begde, Principal Investigator, Loughborough University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5832
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Older People
Keywords: Balance; cognition; exergame; dual-task; older adults

STUDY DESIGN:
Intervention Model Description: Non-randomised controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive dual task training (CDT) Group (Experimental): The CDT group (n = 20) will participate in games on Xbox one consoles that require a higher cognitive demand compared to those of the BDT group. The training sessions will include five different games that require participants to stand and use their hand reach function to interact with different cognitive (i.e. dual-tasking) skills, such as working memory, problem solving, Stroop effect, planning, attention and response time.
  Interventions: Device: Exergame home training programme
- Balance dual task (BDT) training Group (Active Comparator): The BDT group (n = 20) will participate in the conventional training programme on Wii consoles that have been used by previous studies (Barcala et al. 2013; Chao et al. 2015; Kannan et al. 2019), to improve balance performance. The training sessions will include five different games that require participants to stand and use their weight shift to control the game while maintaining balance.
  Interventions: Device: Exergame home training programme

INTERVENTIONS:
Device: Exergame home training programme — Each training programme (Xbox or Wii Fit) is aimed at improving the following issues: improper weight shifting and reduced dual tasking. The participants will be guided in the first sessions to familiarize themselves with the exercises. Then, they will be allowed to exercise independently at home. Allowing enough practice time before collecting data helps minimize practice effects. practice effects are confounding factors that can affect the results and make it difficult to identify whether the improvement in outcome is due to the training or not. The duration of the training programme will be approximately 30 minutes. Each game will be played three times (the duration for each game is approximately one minute).

SUMMARY:
Balance stability requires both motor and cognitive (mental) functions working together. Balance stability may decrease when performing two tasks at the same time (dual task), as cognitive and motor tasks compete for performing a higher task. Meanwhile, social distance and remote working become a necessity due to Covid-19. The primary aim is to evaluate the feasibility of cognitive exergame training in reducing dual-task costs and improve the balance performance among individuals between 65 and 85 years. The secondary aim is to observe the effectiveness of virtual home exercise on adherence and interactive rate of the population between 65 and 85 years.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 65-85 years
* Individuals with no sign of aphasia
* Individuals with a manual muscle test score of ≤5/5
* Individuals who can perform a full range of movement (ROM) against gravity
* Individuals who can stand for five minutes without the use of an assistive device

Exclusion Criteria:

* Individuals with a neurological condition (e.g. vestibular deficit, stroke, Parkinson's disease, epilepsy or peripheral neuropathy) o Individuals with a cardiovascular or musculoskeletal disorder
* Individuals with any lower limb injury or balance disorder within the last 12 months that has affected their physical activity
* Individuals with cognitive impairment such as dementia
* Individuals who score over 13 points on the Short FES-I

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dual-task cost | 8 weeks
  A dual-task cost (DTC) occurs when attention is divided between two tasks (e.g. cognitive and motor tasks), or a delay in one task causes attention to divert to the other. This may cause a decline in balance stability and an increase in dual-task cost. Calculation of dual-task cost A decrease in dual-task performance (i.e. dual-task cost) is represented with a negative value, whereas an improvement in dual-task performance is represented by a positive value.
  DTE(%)=((dual task - single task))/(single task )× 100% An example of the formula for measuring dual-task interference using absolute values of LOS parameters is DTE(%)=((dual-task LOS (RT) - single task LOS (RT)))/(single task LOS (RT)) × 100% An increase in response latency indicates a reduction in performance, thus the following will be used instead: DTE(%)=(-(dual task - single task))/(single task )× 100%
Change in Static balance task | 8 weeks
  The static balance is the ability to keep standing steady with eyes open and with eyes closed without losing balance or taking a step (Winter 1995). The following centre of pressure COP parameters will be computed separately for the anteroposterior (AP) and Mediolateral (ML) directions, such The COP mean velocity (MV), stander deviation (SD) and total displacement area (TD) parameters.

SECONDARY OUTCOMES:
Change in Limit of stability task | 8 weeks
  Limit of stability (LOS) is the amount of the maximum excursion of COP that can be achieved within the supported base without losing balance or taking a step. The dependent variable for LOS is COP parameters that will be collected separately for the (AP) and (ML) directions, such as the COP mean velocity, COP path and COP range (Juras et al. 2008).
Change in Arithmetic tasks | 8 weeks
  Arithmetic cognitive tasks will be measured using the parameters of response latency and response accuracy. Response latency is defined as 'the time from stimulus onset to response onset', and response accuracy is defined as 'the number of correct responses divided by the total number of responses, expressed as a percentage. The cognitive task will only record at 80% of the correct responses or higher. This technique can help to identify if the cognitive task provides an adequate challenge for participants and minimize any learning effect.
Change in Functional Reach (FR) Test | 8 weeks
  FR will measure the maximal distance that can be reached forward beyond the arm's length, without moving the feet. A yardstick will be used to measure the forward reaching length in (cm).
Change in Visual sensitivity test | 8 weeks
  The computerized visual search and detection test requires the disengagement from one focal area of attention to locate the next target (a triangle formed from constantly moving dots). The participant is instructed to press a key as soon as they could detect a triangle on the screen. The baseline level contained 15 stimuli, which are drawn in solid green lines on a black background. In the 40 complex-level stimuli, moving random dots covering the entire screen serve as background distractors. New target triangles are initially drawn with just a few visible dots of each line, and the density of these points increased linearly with time until a keypress response is registered. The screen is redrawn every 250 ms. After each response, new targets appear with random delays of at least 500 ms. Visual search results are recorded with reaction time (in ms) and the number of true and false positives.
Change in Corsi Block-Tapping Test | 8 weeks
  The test is one of the most commonly used tests to measure the visuospatial short-term and working memory. This computerised test consists of nine cubical blocks positioned on the screen. The blocks are tapped in a specific sequence (the colour of tapped blocks change). The participant is asked to remember and tap these blocks in the same sequence. The sequences are easy at the beginning, usually involving three blocks, but they become more difficult in the later stages. The results are recorded with reaction time (in ms) and the number of true and false positives. The test takes around 5 mins.
Change in Hopkins Verbal Learning Test | 8 weeks
  Each form of the Hopkins Verbal Learning Test (HVLT) consists of a 12-item word list of four words from each of the three meaning categories. The participant is instructed to listen carefully as the assessor reads the word list and tries to memorize the words. The word list is then read to the subject at a rate of about one word every 2 seconds. The patient's free recall of the list is recorded. The same procedure is done for two more attempts. After the third learning attempt, the patient is read 24 words and asked to say "yes" after each word (12 goals) that appears on the recall list, and "no" after each word (12 distractors) that does not appear. Half of the distractors are taken from the same semantic categories as the targets (relevant distractors) and a half from other categories (unrelated distractors).
Change in Mobility (Fall Risk) | 8 weeks
  Timed up and go test (<3 min) The participant is asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. The time is recorded.
Change in Stroop Colour-Word test | 8 weeks
  The test measures the sensitivity to interference and the ability to suppress an automated response (time needed to read the colour words rather than the time it takes to name the colour of the letters). The baseline level contains 15 stimuli (reading colour names printed in white on a black background), the colour-interference level (naming the font colour rather than reading the printed colour name, which is always incongruent) comprise 40 stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Begde, Principal Investigator — Loughborough University; Alaa Algurafi, Principal Investigator — Loughborough University; Matthew Pain, Study Director — Loughborough University; Glen Blenkinsop, Study Director — Loughborough University; Eef Hogervorst, Study Director — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No